CLINICAL TRIAL: NCT05945303
Title: Correlation Between Internal Jugular Vein Ultrasound and Electrical Cardiometry in Assessment of Fluid Responsiveness in Patients Undergoing Coronary Artery Bypass Grafting Surgery
Brief Title: Correlation Between Internal Jugular Vein Ultrasound and Electrical Cardiometry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Anas Ezzat Fathy
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Coronary Bypass Stenosis; Coronary Artery Bypass Grafting Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Responder group (Experimental): About 20 Adult patients Planned for elective CABG surgery
  Interventions: Procedure: Coronary Artery Bypass Grafting surgery
- Not Responder group (Experimental): About 20 Adult patients Planned for elective CABG surgery
  Interventions: Procedure: Coronary Artery Bypass Grafting surgery

INTERVENTIONS:
Procedure: Coronary Artery Bypass Grafting surgery — Assessing the reliability of predicting fluid responsiveness in adults undergoing coronary artery bypass graft surgery using ultrasonography of the internal jugular vein for assessment of vessel distensibilty in relation to stroke volume variation (SVV) measured by electrical cardiometry.

SUMMARY:
Coronary artery bypass graft (CABG) surgery is one of the most frequently performed cardiac surgery procedures worldwide. CABG has been used for more than 40 years to relieve symptoms and to reduce the risk of death in patients with ischemic heart disease.

DETAILED DESCRIPTION:
Cardiopulmonary bypass can produce changes in fluid physiology and fluid responsiveness in patients characterized by increased interstitial fluid as a consequence of decreased cardiac output and inflammatory changes. This shift of fluid from intravascular space to the intrtstitial space, in addition to blood and fluid losses during the surgical procedure can result in an intravascular hypovolemia that requires fluid resuscitation.

Fluid management is one of the most important treatments for stabilizing hemodynamics in patients during and after cardiac surgery. Hypovolemia may leads to inadequate organ perfusion, whereas fluid overload may lead to postoperative complications such as congestive heart failure or pulmonary edema, In addition to patients who underwent cardiac surgery have a certain degree of myocardial stunning and hence cautions should be taken regarding fluid management in patients with limited cardiac reserve.

Fluid responsiveness (FR) is generally defined as an increase of 10-15% in stroke volume (SV), cardiac output (CO), or cardiac index (CI) in response to volume expansion and indicates unmasked hypovolemia or preload dependacy.

The methods for assessing fluid responsiveness have been evolved from static and volume parameters such as central venous pressure (CVP), pulmonary artery occlusion pressure (PAOP), inferior vena cava (IVC) and superior vena cava (SVC) diameters, right ventricular end-diastolic volume and right ventricular end-diastolic volume, which are unable to predict fluid responsiveness to dynamic indices such as pulse pressure variation (PPV),stroke volume variation (SVV), Pleth variability index (PVI) and aortic blood flow which is based on heart-lung interactions during mechanical ventilation, which have amodest degree of accuracy.

Techniques based on either a virtual or real fluid challenge such as passive led raising (PLR) and rapid fluid challenge (100-250cc) have a high degree of accuracy in predicting fluid responsiveness.

Over the last decade, a number of studies have used heart-lung interactions during mechanical ventilation to assess fluid responsiveness; specifically pulse pressuer variation (PPV) derived from analysis of the arterial blood pressure wave form, stroke volume variation (SVV) derived from pulse-contour analysis (measured by lithium dilution cardiac output monitoring system (LiDDCO) or pulse index continuous cardiac output monitoring system (PiCCO), and the variation of the amplitude of the pulse oximter plethysmographic waveform have been shown to be highly predictive of fluid responsiveness.

However, dynamic parameters are unreliable during spontaneous breathing activity. To overcome the limited accuracy of these hemodynamic parameters in this specific clinical scenario, a passive leg raising (PLR) manoeuver has been suggested to be reliable predictor of fluid responsiveness during spontaneous breathing.

SVV can be monitored with the PiCCO system requiring transpulmonary thermodilution,It is an invasive procedure requires the venous access and balloon flotation of the catheter through the right side.

Accordingly, there are complications associated with detection with this system, and some are even fatal. Furthermore, this system requires an elaborate protocol for intermittent injections into pulmonary artery catheter thermodilution.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (above 18 years old to be able to provide advanced informed consent Planned for elective CABG surgery) both male and female will be included in the study

Exclusion Criteria:

* Severely reduced preoperative left ventricular ejection fraction (< 40 %).
* Patients who will develop any complication after fluid infusion as pulmonary edema and heart failure will be excluded from the study.
* Significant cardiac arrhythmia.
* Significant valvular heart disease.
* Clinically evident pulmonary disease.
* Bilaterally inserted venous catheters (jugular or subclavian vein).
* History of radiotherapy or surgery of the neck region.
* Inability to obtain interpretable ultrasound images due to a difficult acoustic window.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Reliability of predicting fluid responsiveness | 2 hours after the coronary artery bypass graft surgery
  to assess the reliability of predicting fluid responsiveness in adults undergoing coronary artery bypass graft surgery using ultrasonography of the internal jugular vein for assessment of vessel distensibilty in relation to stroke volume variation (SVV) measured by electrical cardiometry.

SECONDARY OUTCOMES:
Thoracic fluid content | 2 hours after the coronary artery bypass graft surgery
  Evaluate the ability of thoracic fluid content (TFC) measured by electrical cardiometry to be an additive for the assessment of fluid responsiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Mofeed Abdallah, Professor, Study Chair — Al-Azhar University, Faculty of medicine for boys; Mohamed Abdelgawad, Assist.Professor, Study Director — Department of Anesthesia,Faculty of Medicine,Al-Azhar University
Locations (1):
- Al-Azhar University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided